CLINICAL TRIAL: NCT03306186
Title: Integration of Clinical and Laboratory Information to Generate Technological Advance for the Diagnosis of Sepsis
Brief Title: Hemospec Device for the Diagnosis of Sepsis
Acronym: INTELLIGENCE-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Collaborators: Ippokration General Hospital (Other); Tzanion General Hospital of Piraeus (Unknown); Aghia Olga Konstantopouleion General Hospital (Unknown)
Responsible Party: Principal Investigator, Evangelos J. Giamarellos-Bourboulis, M.D., Associate Professor of Internal Medicine, University of Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: INTELLIGENCE1
Record Dates: First submitted 2017-10-03; First posted 2017-10-10 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Sepsis
Keywords: diagnosis; prognosis
MeSH Terms: conditions — Sepsis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HemoSpec (Experimental): Diagnosis of sepsis using HemoSpec device
  Interventions: Device: HemoSpec

INTERVENTIONS:
Device: HemoSpec — Blood sampling for analysis

SUMMARY:
A diagnostic devise, namely HemoSpec, had been developed that integrates clinical information, along with information on circulating protein biomarkers and the morphology of white blood cells to achieve early diagnosis of sepsis. The current study is aiming to validate and improve performance of HemoSpec for the rapid assessment of the critically ill patient.

DETAILED DESCRIPTION:
Sepsis is a life-threating organ dysfunction resulting from the dysregulated response of the host to an infection. It is estimated that 1.5 million people present with sepsis annually in Northern America and another 1.5 million people in Europe; 30 to 50% of them die making sepsis the leading cause of death. The key-point in the management of sepsis is the early resuscitation with broad-spectrum antimicrobials and intravenous fluids, if possible within the first hour. The great mortality of sepsis indicates that this goal is not easy to be achieved for two main reasons: the first is the delay in recognition of the septic patients and the second is the resistance of the implicated pathogen to broad-spectrum antimicrobials.

In an attempt to improve the failure of physicians for early sepsis recognition, several markers have been developed. Some of them rely on clinical signs of the host and others on the measurements of circulating biomarkers. Recently, qSOFA (quick SOFA score) has been introduced to help the early recognition of sepsis in patients who present with infection outside the Intensive care Unit (ICU) i.e. either in the community or during hospitalization in the general ward1. However, there are concerns of the sensitivity of qSOFA and many introduce the need to measure biomarkers in serum. These biomarkers are usually protein molecules that are over-produced in the host as a result of the interaction with an infective insult. However, these protein molecules are produced by white blood cells. What is currently known is that although most of patients present with a similar phenotype, their pathophysiology is diverse. More precisely, although the majority of patients with sepsis present with high concentrations of protein molecules like interleukin (IL)-6, C-reactive protein (CRP) and procalcitonin (PCT) in their blood, in some patients circulating white blood cells remain over-active and in other patients they are significantly anergic, a situation often known as sepsis-induced immunoparalysis. Another molecule, called soluble urokinase plasminogen activator receptor (suPAR), is the shed uPAR receptor on neutrophils and is released in the circulation as a result of neutrophil activation; concentrations greater than 12 ng/ml can trace with negative predictive value almost 95% the patient at great chance of unfavorable outcome. As such, the robust diagnosis of sepsis may rely on a combination of clinical assessment, measurement of protein biomarkers and validation of the activity of circulating white blood cells.

One FrameWork 7-funded initiative from seven European countries aims to develop a rapid score that can integrate all clinical and laboratory information and provide early diagnosis whether a patient has sepsis or not. The vision of this initiative is to build a device that is called HemoSpec. With this approach, whole blood coming from patients will be in parallel analyzed into three aspects: a) absolute white blood cell counting; b) information on the fluidity and activity of the white blood cells using Raman spectroscopy; and c) measurement of serum levels of IL-6, CRP, PCT and suPAR. The end result is building a diagnostic algorithm where clinical information is also taken into consideration.

The project was started in November 2013 and the HemoSpec device is anticipated to be ready by February 2017. The diagnostic performance of HemoSpec is currently based on preliminary data coming from 60 patients (20 controls, 20 with systemic inflammatory response syndrome and 20 with sepsis) hospitalized in Jena University Hospital. The current study is aiming to validate and improve performance of HemoSpec for the rapid assessment of the critically ill patient in a larger phase II diagnostic study.

ELIGIBILITY:
Inclusion Criteria:

* Age above or equal to 18 years old
* Both genders
* Written consent provided from patients or their first-degree relatives for patients unable to consent
* Patients with acute pancreatitis or post-operative or with clinical signs of infection
* Considerable risk of death as as indicated by the presence of at least one of the following: i) sudden alteration of mental status; ii) systolic blood pressure less than 100 mmHg; and iii) high respiratory rate defined as more than or equal to 22 breaths per minute.

Exclusion Criteria:

* Known infection by the human immunodeficiency virus-1;
* Neutropenia defined as an absolute neutrophil count lower than 1000 neutrophils/mm3 due to reasons other than an infection.
* Single trauma or multiple injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity of HemoSpec for the diagnosis of sepsis | 3 days
  The sensitivity of HemoSpec output to diagnose the presence of sepsis compared to the absence of sepsis. HemoSpec output will be considered to provide a satisfactory diagnosis of sepsis if sensitivity for the diagnosis is greater than 85%.

SECONDARY OUTCOMES:
Diagnostic performance for sepsis | 3 days
  The diagnostic performance of HemoSpec output to diagnose the presence of sepsis compared to the absence of sepsis. The diagnostic performance is composed by the aggregation of specificity, positive predictive value and negative predictive value.
Prognostics performance for sepsis | 28 days
  The prognostic performance of HemoSpec output to predict unfavorable outcome compared to survivors. The prognostic performance is composed by the aggregation of sensitivity, specificity, positive predictive value and negative predictive value.
Prognostic performance for organ dysfunction | 28 days
  The prognostic performance of HemoSpec output to predict progression into organ dysfunction. The prognostic performance is composed by the aggregation of sensitivity, specificity, positive predictive value and negative predictive value.
Diagnostic performance over qSOFA | 3 days
  The aggregation of sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of HemoSpec output to indicate patients with infection among those scoring positive for qSOFA.
Diagnostic performance and microbiology | 3 days
  The diagnostic performance of HemoSpec output to diagnose the presence of sepsis between patients with microbiologically-proven infection and patients without microbiologically-proven infection. The diagnostic performance is composed by the aggregation of sensitivity, specificity, positive predictive value and negative predictive value.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos J Giamarellos-Bourboulis, MD, PhD, Study Chair — National and Kapodistrian University of Athens; Konstantinos Toutouzas, MD, PhD, Principal Investigator — National and Kapodistrian University of Athens; Athanasios Prekates, MD, PhD, Principal Investigator — Tzaneion General Hospital; Stylianos Karatzas, MD, PhD, Principal Investigator — Ippokration General Hospital; Christos Mathas, MD, Principal Investigator — Aghia Olga General Hospital
Locations (5):
- Greece (5):
  - 1st Department of Propedeutic Surgery, Ippokration General Hospital, Athens
  - Intensive Care Unit, Ippokration General Hospital, Athens
  - 4th Department of Internal Medicine, ATTIKON University Hospital, Athens
  - Intensive Care Unit, Aghia Olga Konstantopouleion General Hospital, Athens
  - Intensive Care Unit, Tzanio Hospital of Piraeus, Piraeus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Becker KL, Snider R, Nylen ES. Procalcitonin assay in systemic inflammation, infection, and sepsis: clinical utility and limitations. Crit Care Med. 2008 Mar;36(3):941-52. doi: 10.1097/CCM.0B013E318165BABB. PMID 18431284
- [Background] Giamarellos-Bourboulis EJ, Norrby-Teglund A, Mylona V, Savva A, Tsangaris I, Dimopoulou I, Mouktaroudi M, Raftogiannis M, Georgitsi M, Linner A, Adamis G, Antonopoulou A, Apostolidou E, Chrisofos M, Katsenos C, Koutelidakis I, Kotzampassi K, Koratzanis G, Koupetori M, Kritselis I, Lymberopoulou K, Mandragos K, Marioli A, Sunden-Cullberg J, Mega A, Prekates A, Routsi C, Gogos C, Treutiger CJ, Armaganidis A, Dimopoulos G. Risk assessment in sepsis: a new prognostication rule by APACHE II score and serum soluble urokinase plasminogen activator receptor. Crit Care. 2012 Aug 8;16(4):R149. doi: 10.1186/cc11463. PMID 22873681